CLINICAL TRIAL: NCT01612208
Title: Healing of Distal Femur Fractures Stabilized With a Flexible Plating Construct Using MotionLoc Screws
Brief Title: MotionLoc Study, Femur Fractures
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Legacy Health System (Other)
Responsible Party: Principal Investigator, Eric Kubiak, M.D., University of Utah
Other Study IDs: 51842
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Fracture of the Distal Femur

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Distal femur fractures: (AO/OTA types 33-A and 33-C)
  Interventions: Device: Periarticular Locking Plate (NCB, Zimmer); Device: MotionLoc Screw

INTERVENTIONS:
Device: Periarticular Locking Plate (NCB, Zimmer) — The proximal plate segment will be applied to the diaphysis using four 5.0 mm MotionLoc screws. The plate will not be compressed onto the femoral diaphysis to preserve periosteal perfusion and to enable controlled motion between the plate and the diaphysis. If desirable, temporary spacers of the NCB set may be used in the proximal plate segment to facilitate 1-2 mm plate elevation over the diaphysis. Only MotionLoc screws will be used for fixation of the NCB plate proximal to the fracture site.
Device: MotionLoc Screw — The NCB Polyaxial Locking Plate System is indicated for temporary internal fixation and stabilization of fractures and osteotomies of long bones. These MotionLoc screws have a reduced 3.4 mm diameter mid-shaft section to bypass the near cortex. By avoiding rigid constraint in the near cortex, the MotionLoc screw design increases the working length of the screw, allowing for elastic flexion of the screw shaft within a controlled motion envelope in the near cortex.

SUMMARY:
The objective of this study is to document callus formation and healing of fractures stabilized with locking plates utilizing modern MotionLoc screws that provide controlled axial micro-motion to actively promote fracture healing.

DETAILED DESCRIPTION:
Rigid locked plating constructs can suppress fracture healing, particularly at the near cortex adjacent to the plate where interfragmentary motion is minimal. Dynamic fixation with Far Cortical Locking (FCL) screws reduces construct stiffness and induces axial interfragmentary motion to stimulate symmetric callus formation and healing. Two versions of FCL screws are commercially available, but the clinical durability of this novel concept has not been documented to date. This prospective observational study documented our early clinical experience with MotionLoc® FCL screws for stabilization of distal femur fractures to assess their durability and potential complications.

Thirty-two consecutive patients with 33 distal femur fractures (AO/OTA types 33-A and 33-C) were prospectively enrolled at three trauma centers. Fractures were stabilized by plate osteosynthesis with MotionLoc® FCL screws without supplemental bone graft or bone morphogenic proteins. Thirty patients with 31 fractures were available for follow-up until union or revision. Follow-up visits at 6, 12, and 24 weeks comprised functional and radiographic assessment of implant fixation and fracture healing, including computed tomography scans at week 12. The primary endpoint was fracture healing in absence of complications and revision.

There was no incidence of implant breakage or diaphyseal fixation failure. Thirty of 31 fractures healed within 15.6 ± 6.2 weeks, as evident by bridging callus and pain-free load bearing. There were two revisions, one at 5 days post surgery to correct a mal-rotation, and one at 6 months post surgery to revise a non-union. Periosteal callus distribution at week 6 was symmetrical, with similar amounts of callus at the medial cortex (35%) anterior cortex (30%) and posterior cortex (35%). In 23 fractures (74%), callus formation extended to the lateral cortex under the plate.

Absence of hardware and fixation failure suggests that dynamic plating of distal femur fractures with FCL screws provides safe and effective fixation. Moreover, the amount and symmetric distribution of periosteal callus suggests that dynamic fixation with FCL screws may promote increased fracture healing over standard locked plating. However, this hypothesis on the stimulatory effect of dynamic fixation on fracture healing requires investigation in a future randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal femur fracture (AO/OTA Type 33A and 33C).
* Patients 17 years of age and older.
* Patients able to be operated on by selected surgeons at the participating centers.

Exclusion Criteria:

* Pregnancy
* Patients who are enrolled in an investigational treatment trial.
* Patients who are not expected to survive the follow-up period.
* Considered an inappropriate participant by the study physician.
* Revision surgery.
* Patients currently incarcerated or awaiting incarceration.
* Severe spinal injury with neurological deficit resulting in paralysis.
* Fracture fixed more than 28 days after injury.
* Acute or chronic of systematic infections
* Patients with periprosthetic fractures.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Distal femur fractures (AO/OTA Type 33A and 33C)
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Fracture Healing | 6, 12, and 24 weeks post surgery
  Fracture healing is defined clinically by the ability of pain-free weight bearing, and radiographically by callus formation and bridging.

SECONDARY OUTCOMES:
Periosteal Callus Size | 6, 12, 24 weeks post surgery
  Periosteal callus size is assessed at the anterior, posterior, and medial aspects on radiographs using a validated computational algorithm.
Bridging Callus from CT | 12 weeks post surgery
  Cross-sectional image analysis, supported by 3-D rendering, to detect bony bridging at the anterior, posterior, and lateral aspects of the femur.
Fixation Failure | 24 weeks post surgery
  Assessed in terms of loss of alignment at 12 and 24 weeks post surgery
Hardware failure | 6, 12, 24 weeks post surgery
  Breakage of screw or plate

CONTACTS AND LOCATIONS:
Overall Officials: Erik Kubiak, Principal Investigator — Orthopedic Surgery Operations